CLINICAL TRIAL: NCT06456333
Title: Paravertebral Electromyographic Characteristics of Adolescent Idiopathic Scoliosis Patients Explored on the Basis of High-density Surface Electromyography
Brief Title: Exploring Paraspinal Electromyographic Features in Adolescent Idiopathic Scoliosis Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-K-286-01
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Scoliosis; Adolescence; Electromyography
Keywords: Adolescent idiopathic scoliosis; high-density surface electromyography; Cross-sectional study
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescent idiopathic scoliosis patients（Observation Group）: Acquisition equipment：SAGA high-density electromyography system (TMSi, New Zealand).Acquisition site: paravertebral muscle at the L1-L3 level, with the electrode sheet placed 1.5 cm adjacent to the spinous process.Acquisition process: ① Place the electrode sheet and fix it. ② The subject was instructed to complete the specified movements according to the experimental paradigm and the EMG signals were recorded simultaneously.Experimental Paradigm:Biering-Sorensen test,BST：The subject was lying prone on the bed, with the upper half of the body poking out of the bed, the anterior superior iliac spine located at the edge of the bed, both lower limbs partially immobilized on the bed with straps, both hands crossed in front of the chest grasping the contralateral shoulder and tightly pressed against the chest wall, and the torso was suspended in the air and parallel to the floor, and the patient stopped the test when he/she maintained this position for 90s.
  Interventions: Device: High-density surface electromyography
- Healthy population（Control Group）: Same intervention as the observation group.
  Interventions: Device: High-density surface electromyography

INTERVENTIONS:
Device: High-density surface electromyography — Electromyographic signals were acquired from the paravertebral muscles in apical vertebral in patients with AIS using SAGA High Density Myoelectrics (TMSi International, New Zealand)

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a complex three-dimensional spinal deformity with onset in adolescents between the ages of 10 and 18 years, characterized by coronal curvature, sagittal imbalance and horizontal rotation of the spine. The incidence of AIS is 1-4% globally, with more females than males, and it is a common, frequent and difficult-to-treat disease that seriously jeopardizes the physical and mental health of adolescents.

Previous studies have found significant changes in the morphologic structure and physiologic characteristics of the paraspinal muscles in patients with AIS, including muscle fiber distribution, muscle contraction and relaxation capacity, the convex side of the AIS curve exhibits a higher level of electromyographic activity, and asymmetric changes in the paraspinal muscles are highly correlated with progression of scoliosis. The current single-electrode sEMG technique extracts limited muscle activity signals and is susceptible to interference from random noise. Compared with the single-electrode sEMG technique, HD-sEMG can provide rich spatiotemporal information on paraspinal muscle activity, so it is necessary to use a wide and closely spaced electrode array for signal acquisition to obtain more accurate and detailed characteristics of paraspinal muscle activity.

In summary, this study used high-density surface electromyography to collect muscle parameters of the paraspinal muscles on the concave and convex sides of AIS patients and compared them with those of healthy people to comprehensively summarize the characteristics of their paraspinal muscles, so as to provide scientific basis for the subsequent development of precise treatment plans and improvement of clinical efficacy.

DETAILED DESCRIPTION:
Paravertebral muscle EMG signals were acquired from AIS patients and healthy controls under the BST test paradigm.

Acquisition site: paravertebral muscle at the L1-L3 level, with the electrode sheet placed 1.5 cm adjacent to the spinous process.

（Biering-Sorensen test,BST）：The subject was lying prone on the bed, with the upper half of the body poking out of the bed, the anterior superior iliac spine located at the edge of the bed, both lower limbs partially immobilized on the bed with straps, both hands crossed in front of the chest grasping the contralateral shoulder and tightly pressed against the chest wall, and the torso was suspended in the air and parallel to the floor, and the patient stopped the test when he/she maintained this position for 90s.

Observation indicators:

1, the average change (mean) characteristics of each channel signal, including the 32 channels of the root mean square value （RMS）, mean power frequncy（MPF）, fractal dimension（FD）,Slope sign change(SSC), a total of 4 types of indicators-reflecting the strength and fatigue of muscle contractions..

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AIS
* Any gender, age 10-18 years old
* Signed informed consent and able to cooperate with follow-up
* Ability to cooperate with electromyography examination and evaluation, and to perform measurements of relevant indexes.

Exclusion Criteria:

* Subjects with spine-related diseases such as Marfan's syndrome
* Subjects with previous spine-related diseases such as ankylosing spondylitis, spinal neurofibroma, spinal tuberculosis, spinal trauma, etc
* Subjects with comorbid serious medical diseases and patients with psychiatric disorders
* Subjects with ECOG scores of >2, which may have an effect on the results of the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: AIS patients and healthy control populations
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
root mean square value （RMS） | Day 1
  The square root of the mean value of the amplitude of the sEMG signal over a certain time window is commonly used to assess the strength of muscle contraction and fatigue.
mean power frequncy（MPF） | Day 1
  The average of the power frequency distribution of the sEMG signals generated during a muscle contraction can be used to assess the force and fatigue of a muscle contraction.
fractal dimension（FD） | Day 1
  The complex waveforms were categorized into multiple dimensions, and each dimension was analyzed by typing.
Slope sign change(SSC) | Day 1
  The number of times the sign of the rate of change of amplitude changes in the waveform of the sEMG signal is commonly used to indicate an impending fluctuating change in the state of the surface EMG signal.

CONTACTS AND LOCATIONS:
Overall Officials: Honggen Du, doctor, Study Director — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

DOCUMENTS (1):
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT06456333/ICF_000.pdf